CLINICAL TRIAL: NCT01744158
Title: Exploring Hypertonia in Children With Cerebral Palsy- a Population-based Approach.
Brief Title: Exploring Hypertonia in Children With Cerebral Palsy
Acronym: HypE-CP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Women's and Children's Hospital, Australia (Other Government)
Collaborators: Allergan Australia Pty Ltd (Industry)
Responsible Party: Principal Investigator, Dr James Rice, Senior Consultant in Rehabilitation Medicine, Women's and Children's Hospital, Australia
Other Study IDs: REC2202/8/12
Record Dates: First submitted 2012-08-21; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Cerebral Palsy.
Keywords: cerebral palsy; spasticity; dystonia; hypertonia; register; motor function
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Dystonia; Muscle Hypertonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with cerebral palsy: No intervention applicable
  Interventions: Other: No intervention applicable

INTERVENTIONS:
Other: No intervention applicable — Following consent, children will undergo a comprehensive assessment performed by a research team including rehabilitation paediatrician and therapist. Hypertonia and abnormal movements will be assessed by a pediatrician with expertise in treating children with movement disorders. The assessments will be performed at a rehabilitation clinic, or child's home, and will include:
  * differentiation of hypertonia by application of the Hypertonia Assessment Tool-Discriminate (HAT-D)
  * measurement of severity of dystonia using the Barry Albright dystonia scale, based on video recording
  * measurement of severity of spasticity using the modified Ashworth score
  * description of presence of chorea or athetosis
  * classification of gross motor abilities using the GMFCS and functional mobility scale (FMS)
  * classification of fine motor abilities using the manual ability classification system (MACS)
  * collection of demographic data and associated medical history

SUMMARY:
Abnormal limb and trunk movements are seen in many children with cerebral palsy. Recognizing the difference between types of these movements is not well understood. This study aims to describe how common are these movements in children recruited from a population-based sample of children identified on a cerebral palsy register, and to explore associations with motor abilities. It is hoped this will lead to improved understanding and recognition of movement disorders in CP, to allow clinicians to choose appropriate treatments. We hypothesise that the underlying prevalence of dyskinesia is higher than that previously identified through conventional motor descriptions in cerebral palsy populations in Australia, and may approach 20%.

DETAILED DESCRIPTION:
A key descriptor associated with the term cerebral palsy is "the disordered development of movement and posture, resulting in activity limitation." The term "movement disorders" is now commonly used to describe a range of observed abnormal movements and postures displayed by children with chronic neurological conditions, of which cerebral palsy (CP) is the most common. These children have muscle tone abnormalities related to non-progressive damage to motor pathways, in particular those contained within the cortex, basal ganglia and thalamus. In recent years there has been much focus on understanding and treating abnormal tone and movements in children with CP, including spasticity and dystonia. Spasticity, which occurs in approximately 90% of children with CP is defined as the velocity-dependent resistance of a muscle to stretch. In general, spasticity is elicited during a standard clinical examination, such as by passive range of joint motion performed at varying speeds.

Dystonia in childhood is defined as ''a movement disorder in which involuntary sustained or intermittent muscle contractions cause twisting and repetitive movements, abnormal postures, or both. ''. In contrast to spasticity, dystonia is inherently more difficult to observe and measure, particularly when spasticity co-exists. When classified according to the dominant form of tone abnormality, it accounts for up to 2-15% of cases. However it is often overlooked in the diagnostic formulation of motor aspects of cerebral palsy, and therefore does not necessarily figure in treatment decision-making. Under-recognised dystonia, when co-existent with spasticity, can produce unpredictable surgical outcomes in the management of gait disorders and associated musculoskeletal deformities. In addition, other abnormal movements such as chorea and athetosis may be observed in these children, adding to the complexity of the movement disorder, but are rarely classified as dominant abnormalities. Improving the recognition of dyskinesias, and situations where they co-exist with spasticity, is important not only for promoting a clearer description of tone and movement abnormalities, but also to help tailor appropriate treatments leading to improved outcomes.

In our recent study describing the motor profiles of 247 5-year-old children in the South Australian CP population, 93.2% of children were coded as primarily spastic-type; 3.2% as dyskinetic (dystonia or athetosis) and 3.6% as ataxic.1 However this study also found that when children were assessed face-to-face by a group of expert paediatricians, 19.4% of the population was noted on observation alone to have abnormal movements, which included dyskinesias. This increased with motor severity by Gross Motor Functional Classification System (GMFCS) from 7% (level I) to 45% (level V). We questioned whether in fact recognition of some dyskinesias are "masked" by the presence of spasticity, according to conventional clinical descriptors. We advocated for the development of a classification system that describes spasticity and dystonia in parallel, to aid the clinician in prescribing treatment strategies. To date no published study has systematically examined for the prevalence of abnormal movements in CP populations, beyond determining the dominant form of tone abnormality in a mutually exclusive fashion, e.g. spasticity or dystonia. Our study proposes a mutually inclusive format using a recently validated tool for the recognition of dystonia and other abnormal movements.

ELIGIBILITY:
Inclusion Criteria:

* children with a confirmed diagnosis of cerebral palsy
* aged between 2 and 18 years

Exclusion Criteria:

* presence of any progressive neurological disorder, including forms of genetic dystonia
* children less than two years, or greater than 18 years of age

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be those with cerebral palsy attending Rehabilitation clinics at the Women's and Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Hypertonia Assessment Tool-Discriminate (HAT-D) | One hour
  The Hypertonia Assessment Tool (HAT) is a seven-item standardised clinical assessment tool used to differentiate the various types of paediatric hypertonia. There are 2 spasticity items, 2 rigidity items and 3 dystonia items and a standardized protocol for administration has been developed. Each item is scored yes or no. A positive score for at least one item of the subgroup confirms the presence of the subtype of hypertonia in the limb examined.
Barry-Albright Dystonia scale | One hour
  The Barry-Albright Dystonia scale is a 5-point criterion-based ordinal scale for measuring dystonia in CP, with sound validity and reliability. 7 It assesses dystonia in 8 body regions: eyes, mouth, neck, trunk, and the 4 extremities. Severity is scored from none to severe, with each body region having specific descriptors for scoring.

SECONDARY OUTCOMES:
Modified Ashworth Scale | One hour
  The Modified Ashworth scale is a 6-point ordinal scale of muscle tone and involves a subjective assessment of muscle resistance as a limb is moved trough its full passive range.

CONTACTS AND LOCATIONS:
Overall Officials: James E Rice, MD, Principal Investigator — Women's and Children's Health Network
Locations (1):
- Women's and Children's Hospital, Adelaide, South Australia, Australia